CLINICAL TRIAL: NCT01225887
Title: A Phase II Evaluation of BIBF 1120 in the Treatment of Recurrent or Persistent Endometrial Carcinoma
Brief Title: Nintedanib in Treating Patients With Recurrent or Persistent Endometrial Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: GOG Foundation (Network)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GOG-0229K; NCI-2011-02657 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000687306; GOG-DTM0906; GOG-0229K; GOG-0229K (Other: NRG Oncology); GOG-0229K (Other: CTEP); U10CA180868 (NIH); U10CA027469 (NIH)
Record Dates: First submitted 2010-10-20; First posted 2010-10-21 (Estimated); Results first posted 2017-10-09 (Actual); Last update posted 2017-10-09 (Actual); Status verified 2016-10

CONDITIONS: Endometrial Adenocarcinoma; Endometrial Clear Cell Adenocarcinoma; Endometrial Mucinous Adenocarcinoma; Endometrial Serous Adenocarcinoma; Endometrial Squamous Cell Carcinoma; Endometrial Transitional Cell Carcinoma; Endometrial Undifferentiated Carcinoma; Malignant Uterine Corpus Mixed Epithelial and Mesenchymal Neoplasm; Recurrent Uterine Corpus Carcinoma
MeSH Terms: interventions — nintedanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (nintedanib) (Experimental): Patients receive nintedanib PO BID on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Nintedanib

INTERVENTIONS:
Drug: Nintedanib — Given PO
  Other Names: BIBF 1120; BIBF-1120; Intedanib; Multitargeted Tyrosine Kinase Inhibitor BIBF 1120; tyrosine kinase inhibitor BIBF 1120; Vargatef

SUMMARY:
This phase II trial studies the side effects and how well nintedanib works in treating patients with endometrial cancer that has come back. Nintedanib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth or by blocking blood flow to the tumor.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the proportion of patients with persistent or recurrent endometrial cancer, who survive progression-free without going on a subsequent therapy against the disease for at least 6 months and the proportion of patients who have objective tumor response (complete or partial), treated with BIBF 1120 (nintedanib).

II. To determine the nature and degree of toxicity of BIBF 1120 in this cohort of patients.

SECONDARY OBJECTIVES:

I. To estimate the progression-free survival (PFS) and overall survival (OS) of patients with persistent or recurrent endometrial cancer treated with BIBF 1120.

OUTLINE:

Patients receive nintedanib orally (PO) twice daily (BID) on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 2 years and then every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have recurrent or persistent endometrial carcinoma, which is refractory to curative therapy or established treatments; histologic confirmation of the original primary tumor is required; patients with the following histologic epithelial cell types are eligible: endometrioid adenocarcinoma, serous adenocarcinoma, undifferentiated carcinoma, clear cell adenocarcinoma, mixed epithelial carcinoma, adenocarcinoma not otherwise specified (N.O.S.), mucinous adenocarcinoma, squamous cell carcinoma, and transitional cell carcinoma
* All patients must have measurable disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1; measurable disease is defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded); each lesion must be >= 10 mm when measured by computed tomography (CT), magnetic resonance imaging (MRI) or caliper measurement by clinical exam; or >= 20 mm when measured by chest x-ray; lymph nodes must be >= 15 mm in short axis when measured by CT or MRI
* Patient must have at least one "target lesion" to be used to assess response on this protocol as defined by RECIST 1.1; tumors within a previously irradiated field will be designated as "non-target" lesions unless progression is documented or a biopsy is obtained to confirm persistence at least 90 days following completion of radiation therapy
* Patients must not be eligible for a higher priority Gynecologic Oncology Group (GOG) protocol, if one exists; in general, this would refer to any active GOG Phase III protocol or Rare Tumor protocol for the same patient population
* Patients must have a GOG performance status of 0, 1, or 2
* Patients must have normal thyroid function; patients with a history of hypothyroidism are eligible, provided it is well controlled on medication
* Recovery from effects of recent surgery, radiotherapy, or chemotherapy
* Patients should be free of active infection requiring antibiotics (with the exception of uncomplicated urinary tract infection)
* Any hormonal therapy directed at the malignant tumor must be discontinued at least one week prior to registration
* Any other prior therapy directed at the malignant tumor, including chemotherapy and immunologic agents, must be discontinued at least three weeks prior to registration
* Any prior radiation therapy must be completed at least 4 weeks prior to registration
* Patients must have had one prior chemotherapeutic regimen for management of endometrial carcinoma; chemotherapy administered in conjunction with primary radiation as a radio-sensitizer will be counted as a systemic chemotherapy regimen
* Patients are allowed to receive, but are not required to receive, one additional cytotoxic regimen for management of recurrent or persistent disease
* Patients must have NOT received any non-cytotoxic (biologic or targeted) agents, as part of their primary treatment or for management of recurrent or persistent disease; non-cytotoxic (biologic or targeted) agents include (but are not limited to) monoclonal antibodies, cytokines, and small-molecule inhibitors of signal transduction; prior hormonal therapy is allowed; there is no limit on the number of prior hormonal therapies allowed
* Absolute neutrophil count (ANC) greater than or equal to 1,500/mcl
* Platelets greater than or equal to 100,000/mcl
* Creatinine less than or equal to 1.5 x institutional upper limit normal (ULN)
* Urine protein creatinine (UPC) ratio must be < 1.0 gm; if UPC ratio >= 1, collection of 24-hour urine measurement of urine protein is recommended
* Bilirubin must be less than 1.5 X ULN
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) must be less than 3 X ULN
* Alkaline phosphatase must be less than 2.5 X ULN
* Prothrombin time (PT) such that international normalized ratio (INR) is =< 1.5 x ULN (or an in-range INR, usually between 2 and 3, if a patient is on a stable dose of therapeutic warfarin) and a partial thromboplastin time (PTT) =< 1.5 times the institutional upper limit of normal
* Electrocardiogram (EKG) must have corrected QT interval (QTc) < 450 msec without evidence of serious ventricular arrhythmia (ventricular tachycardia lasting more than 3 beats or ventricular fibrillation)
* Patients must have signed an approved informed consent and authorization permitting release of personal health information
* Patients must meet pre-entry requirements
* Patients of childbearing potential must have a negative serum pregnancy test prior to the study entry; women of child-bearing potential must agree to use adequate contraception (two barrier methods of birth control) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she is to inform her treating physician immediately; all patients must be willing to take contraception up to three months after the final dose of BIBF 1120

Exclusion Criteria:

* Patients who have had prior therapy with BIBF 1120
* Patients with a history of other invasive malignancies, with the exception of non-melanoma skin cancer and other specific malignancies, are excluded if there is any evidence of other malignancy being present within the last three years; patients are also excluded if their previous cancer treatment contraindicates this protocol therapy
* Patients who have received prior radiotherapy to any portion of the abdominal cavity or pelvis OTHER THAN for the treatment of endometrial cancer within the last three years are excluded; prior radiation for localized cancer of the breast, head and neck, or skin is permitted, provided that it was completed more than three years prior to registration, and the patient remains free of recurrent or metastatic disease
* Patients who have received prior chemotherapy for any abdominal or pelvic tumor OTHER THAN for the treatment of endometrial cancer within the last three years are excluded; patients may have received prior adjuvant chemotherapy for localized breast cancer, provided that it was completed more than three years prior to registration, and that the patient remains free of recurrent or metastatic disease
* Patients with serious, non-healing wound, ulcer, or bone fracture; this includes history of abdominal fistula, gastrointestinal perforation or intra-abdominal abscess within 28 days prior to the start date of treatment; patients with underlying lesions that caused the fistula or perforation in the past that have not been corrected
* Patients with active bleeding or pathologic conditions that carry high risk of bleeding, such as known bleeding disorder, coagulopathy, or tumor involving major vessels
* Patients with history of brain metastases, or evidence upon physical examination of active central nervous system (CNS) disease, including primary brain tumor, seizures not controlled with standard medical therapy or any brain metastases
* Uncontrolled hypertension, defined as systolic >= 150 mm Hg or diastolic >= 90 mm Hg
* Myocardial infarction or unstable angina within 6 months of study treatment
* New York Heart Association (NYHA) class II or greater congestive heart failure
* Women with an ejection fraction < institutional lower limit of normal (LLN)
* History of serious ventricular arrhythmia (i.e., ventricular tachycardia or ventricular fibrillation) or cardiac arrhythmias requiring anti-arrhythmic medications (except for atrial fibrillation that is well controlled with anti-arrhythmic medication)
* Common Terminology Criteria for Adverse Events (CTCAE) grade 2 or greater peripheral vascular disease
* History of cerebrovascular accident (CVA, stroke), transient ischemic attack (TIA) or subarachnoid hemorrhage within six months of study treatment
* Patients undergoing invasive procedures as defined below: major surgical procedure, open biopsy or significant traumatic injury within 28 days prior to the first date of treatment; major surgical procedure anticipated during the course of the study; minor surgical procedures, fine needle aspirates, or core biopsies within 7 days prior to the first date of therapy
* Patients who are pregnant or nursing
* Patients with a history of major thromboembolic event defined as: symptomatic pulmonary embolism (PE), recurrent asymptomatic PE, or recurrent deep venous thrombosis
* Prior thrombosis or thromboembolic event due to a known inherited coagulopathy (i.e., antithrombin-III deficiency, protein C or protein S deficiency, factor V Leiden mutation presence, prothrombin G20210A mutation)
* Serious infections requiring systemic antibiotics or antiviral therapy including: known active hepatitis B or C infection; known human immunodeficiency virus (HIV) infection
* Gastrointestinal (GI) or other medical disorders that would impact ingestion or absorption of the drug
* Patients with a history of photosensitivity or who must take agents which increase photosensitivity, e.g. topical retinoids and doxycycline
* Patients who are unable to swallow capsules

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2011-10; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Don Dizon, Principal Investigator — NRG Oncology
Locations (59):
- United States (59):
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - University of Colorado Cancer Center - Anschutz Cancer Pavilion, Aurora, Colorado
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - Memorial University Medical Center, Savannah, Georgia
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Northwestern University, Chicago, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Sudarshan K Sharma MD Limted-Gynecologic Oncology, Hinsdale, Illinois
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Saint Vincent Oncology Center, Indianapolis, Indiana
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - MedStar Franklin Square Medical Center/Weinberg Cancer Institute, Baltimore, Maryland
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - Michigan Cancer Research Consortium NCORP, Ann Arbor, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Genesys Regional Medical Center, Grand Blanc, Michigan
  - Allegiance Health, Jackson, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Saint Mary Mercy Hospital, Livonia, Michigan
  - Saint Joseph Mercy Port Huron, Port Huron, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Women's Cancer Center of Nevada, Las Vegas, Nevada
  - Stony Brook University Medical Center, Stony Brook, New York
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Carolinas HealthCare System NorthEast, Concord, North Carolina
  - Akron General Medical Center, Akron, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - Lake University Ireland Cancer Center, Mentor, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - Women and Infants Hospital, Providence, Rhode Island
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Pacific Gynecology Specialists, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Seattle Cancer Care Alliance, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - Northwest Hospital, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
  - Green Bay Oncology at Saint Vincent Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital, Green Bay, Wisconsin
  - Green Bay Oncology Limited at Saint Mary's Hospital, Green Bay, Wisconsin
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Holy Family Memorial Hospital, Manitowoc, Wisconsin
  - Bay Area Medical Center, Marinette, Wisconsin

REFERENCES:
- [Derived] Dizon DS, Sill MW, Schilder JM, McGonigle KF, Rahman Z, Miller DS, Mutch DG, Leslie KK. A phase II evaluation of nintedanib (BIBF-1120) in the treatment of recurrent or persistent endometrial cancer: an NRG Oncology/Gynecologic Oncology Group Study. Gynecol Oncol. 2014 Dec;135(3):441-5. doi: 10.1016/j.ygyno.2014.10.001. Epub 2014 Oct 13. PMID 25312396

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Nintedanib)
Started | 37
Completed | 32
Not Completed | 5
Not completed — Ineligible:required test not done | 2
Not completed — Ineligible;improper pre-protocol therapy | 1
Not completed — Ineligible:inadequate pathology | 2

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Nintedanib)
Number analyzed (Participants) | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.1 (9.8)
Age, Customized [Count of Participants; unit: Participants]
  30-39 years | 1
  50-59 years | 4
  60-69 years | 14
  70-79 years | 10
  80-89 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: The incidence of adverse events (grade 3 or higher) as assessed by the National Cancer Institute CTCAE version 4.0
Time Frame: Up to 5 years
Population: Patients on study who experienced adverse events (Grade 3 or higher)
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Nintedanib)
Number analyzed (Participants) | 32
Participants
  Leukopenia | 1
  Neutropenia | 1
  Anemia | 2
  Other Investigations | 4
  Nausea | 2
  Vomiting | 2
  Other Gastrointestinal | 6
  General & Administration site | 3
  Infections/infestations | 1
  Metabolism/nutrition | 1
  Musculoskeletal/connective tissue | 2
  Psychiatric | 2
  Renal/Urinary | 4
  Respiratory/thoracic/mediastinal | 2
  Vascular Disorders | 1

2. Primary Outcome: Objective Tumor Response
Description: Complete and Partial Tumor Response by RECIST 1.1
Time Frame: For disease that can be evaluated by physical exam,response was assessed prior to each cycle CT scan or MRI if used to follow lesion for measurable disease every other cycle up to 5 years.
Population: Eligible and Treated Patients
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Nintedanib)
Number analyzed (Participants) | 32
percentage of participants | 9.4 [3 to 22]

3. Primary Outcome: Progression-free Survival > 6 Months
Description: Whether or not the patient survived progression-free for at least 6 months.
Time Frame: for disease that can be evaluated by physical exam, progression was assessed prior to each cycle. CT scan or MRI if used to follow lesion for measurable disease every other cycle up to 5 years.
Population: Eligible and Treated Patients
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Nintedanib)
Number analyzed (Participants) | 32
percentage of participants | 21.9 [11 to 37]

4. Secondary Outcome: Overall Survival
Description: The observed length of life from entry into the study to death or the date of last contact.
Time Frame: From study entry to death or last contact, up to 5 years
Population: Eligible and treated patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Nintedanib)
Number analyzed (Participants) | 32
months | 10.1 [5.5 to 14.0]

5. Secondary Outcome: Progression Free Survival
Description: the period of progression free survival for patients with persistent or recurrent endometrial cancer treated with study drug.
Time Frame: The duration of time from study entry to time of progression or death, whichever occurs first, assessed up to 5 years
Population: The time in months that a patient survived progression-free.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Treatment (Nintedanib)
Number analyzed (Participants) | 32
months | 3.3 [1.9 to 3.8]

ADVERSE EVENTS:
Time Frame: All Adverse Events (AEs) occurring during treatment and up to 30 days after stopping the study treatment are reported. Also reported are Serious Adverse Events (SAEs) considered to be treatment related for up to 5 years after stopping study treatment.
Arm/Group | Treatment (Nintedanib)
Serious Adverse Events (participants affected / at risk) | 14/32
Other Adverse Events (participants affected / at risk) | 32/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Nintedanib) (N=32)
Colonic Obstruction (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Ascites (Gastrointestinal disorders) | 1
Jejunal Obstruction (Gastrointestinal disorders) | 1
Fever (General disorders) | 1
Kidney Infection (Infections and infestations) | 1
Aspartate Aminotransferase Increased (Investigations) | 1
Alanine Aminotransferase Increased (Investigations) | 1
Flank Pain (Musculoskeletal and connective tissue disorders) | 1
Urinary Tract Obstruction (Renal and urinary disorders) | 1
Acute Kidney Injury (Renal and urinary disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Thromboembolic Event (Vascular disorders) | 2
Hypertension (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Nintedanib) (N=32)
Anemia (Blood and lymphatic system disorders) | 15
Cardiac Disorders - Other (Cardiac disorders) | 1
Sinus Tachycardia (Cardiac disorders) | 2
Tinnitus (Ear and labyrinth disorders) | 2
Glaucoma (Eye disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Dry Mouth (Gastrointestinal disorders) | 2
Colonic Hemorrhage (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 6
Diarrhea (Gastrointestinal disorders) | 21
Vomiting (Gastrointestinal disorders) | 13
Abdominal Pain (Gastrointestinal disorders) | 13
Rectal Hemorrhage (Gastrointestinal disorders) | 1
Abdominal Distension (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 21
Ascites (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 2
Gastritis (Gastrointestinal disorders) | 1
Pain (General disorders) | 4
Malaise (General disorders) | 1
Non-Cardiac Chest Pain (General disorders) | 1
Edema Limbs (General disorders) | 3
Fatigue (General disorders) | 18
Fever (General disorders) | 1
Portal Vein Thrombosis (Hepatobiliary disorders) | 1
Upper Respiratory Infection (Infections and infestations) | 1
Skin Infection (Infections and infestations) | 1
Esophageal Infection (Infections and infestations) | 1
Urinary Tract Infection (Infections and infestations) | 1
Weight Loss (Investigations) | 4
Platelet Count Decreased (Investigations) | 3
Lymphocyte Count Decreased (Investigations) | 2
Inr Increased (Investigations) | 2
Ggt Increased (Investigations) | 1
Creatinine Increased (Investigations) | 4
Cholesterol High (Investigations) | 1
Neutrophil Count Decreased (Investigations) | 4
Blood Bilirubin Increased (Investigations) | 2
White Blood Cell Decreased (Investigations) | 6
Aspartate Aminotransferase Increased (Investigations) | 13
Alkaline Phosphatase Increased (Investigations) | 11
Alanine Aminotransferase Increased (Investigations) | 13
Hypophosphatemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 4
Hypomagnesemia (Metabolism and nutrition disorders) | 6
Hypokalemia (Metabolism and nutrition disorders) | 7
Hypoglycemia (Metabolism and nutrition disorders) | 1
Hypocalcemia (Metabolism and nutrition disorders) | 4
Hypoalbuminemia (Metabolism and nutrition disorders) | 5
Hyperuricemia (Metabolism and nutrition disorders) | 1
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1
Hypernatremia (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 9
Dehydration (Metabolism and nutrition disorders) | 2
Anorexia (Metabolism and nutrition disorders) | 10
Acidosis (Metabolism and nutrition disorders) | 1
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Generalized Muscle Weakness (Musculoskeletal and connective tissue disorders) | 1
Flank Pain (Musculoskeletal and connective tissue disorders) | 1
Bone Pain (Musculoskeletal and connective tissue disorders) | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 4
Peripheral Sensory Neuropathy (Nervous system disorders) | 5
Memory Impairment (Nervous system disorders) | 1
Headache (Nervous system disorders) | 7
Dysgeusia (Nervous system disorders) | 2
Dizziness (Nervous system disorders) | 2
Insomnia (Psychiatric disorders) | 4
Depression (Psychiatric disorders) | 5
Confusion (Psychiatric disorders) | 1
Anxiety (Psychiatric disorders) | 2
Urinary Urgency (Renal and urinary disorders) | 1
Urinary Frequency (Renal and urinary disorders) | 2
Proteinuria (Renal and urinary disorders) | 1
Hematuria (Renal and urinary disorders) | 5
Acute Kidney Injury (Renal and urinary disorders) | 2
Vaginal Hemorrhage (Reproductive system and breast disorders) | 2
Dyspareunia (Reproductive system and breast disorders) | 1
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 1
Postnasal Drip (Respiratory, thoracic and mediastinal disorders) | 2
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 6
Allergic Rhinitis (Respiratory, thoracic and mediastinal disorders) | 1
Adult Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Skin Hyperpigmentation (Skin and subcutaneous tissue disorders) | 1
Rash Acneiform (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1
Thromboembolic Event (Vascular disorders) | 2
Lymphedema (Vascular disorders) | 1
Hypertension (Vascular disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No